CLINICAL TRIAL: NCT01457469
Title: Adapting Smoking Cessation Interventions for the Outpatient Oncology Setting
Brief Title: Enhanced Quitline Intervention in Smoking Cessation for Patients With Non-Metastatic Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00014657; NCI-2011-02410 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 99310 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2011-10-21; First posted 2011-10-24 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Limited Stage Small Cell Lung Cancer; Recurrent Small Cell Lung Cancer; Stage IA Non-small Cell Lung Cancer; Stage IB Non-small Cell Lung Cancer; Stage IIA Non-small Cell Lung Cancer; Stage IIB Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Tobacco Use Disorder
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Tobacco Use Disorder | interventions — Counseling; Early Intervention, Educational; Methods; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (usual care plus) (closed to accrual as of 3/6/2012) (Active Comparator): Patients receive a personalized letter from their physician with advice to quit smoking and a copy of the National Cancer Institute's "Cleaning the Air" smoking cessation booklet.
  Interventions: Other: questionnaire administration; Procedure: quality-of-life assessment; Other: educational intervention
- Arm II (enhanced quitline) (Experimental): Patients receive a personalized letter and a smoking cessation booklet. Patients also receive an 8-week supply of nicotine replacement patches and undergo a counseling session over 30-45 minutes with a trained nurse or midlevel provider that focuses on the benefits of quitting smoking for cancer patients and addresses cancer-specific concerns about smoking cessation. Patients also undergo a quitline-based smoking cessation intervention comprising 5 individual 25- to 30-minute telephone counseling sessions and unlimited inbound phone-based access to Quit Coaches over 8-11 weeks, mailed written materials, and an interactive online program.
  Interventions: Other: questionnaire administration; Procedure: quality-of-life assessment; Other: counseling intervention; Other: internet-based intervention; Behavioral: telephone-based intervention; Drug: nicotine replacement therapy; Other: educational intervention

INTERVENTIONS:
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: counseling intervention — Undergo counseling session
  Other Names: counseling and communications studies
  Arms: Arm II (enhanced quitline)
Other: internet-based intervention — Receive enhanced quitline intervention
  Arms: Arm II (enhanced quitline)
Behavioral: telephone-based intervention — Receive enhanced quitline intervention
  Arms: Arm II (enhanced quitline)
Other: educational intervention — Receive usual care plus
  Other Names: intervention, educational
  Arms: Arm I (usual care plus) (closed to accrual as of 3/6/2012)
Drug: nicotine replacement therapy — Receive nicotine replacement patches
  Other Names: Nicotine Replacement; NRT
  Arms: Arm II (enhanced quitline)
Other: educational intervention — Receive enhanced quitline intervention
  Other Names: intervention, educational
  Arms: Arm II (enhanced quitline)

SUMMARY:
This randomized clinical trial studies enhanced quitline intervention in smoking cessation for patients with non-metastatic lung cancer. Stop-smoking plans suggested by doctors may help patients with early-stage cancer quit smoking

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate the feasibility of delivering an enhanced quitline-based smoking cessation intervention to lung cancer patients in the outpatient oncology setting.

SECONDARY OBJECTIVES:

I. To gather preliminary outcome data for an enhanced quitline-based smoking cessation intervention adapted to the outpatient oncology setting to support future grant applications.

II. To evaluate change in primary patient reported outcomes, including quality of life (quantified by the Functional Assessment of Cancer Therapy - Lung [FACT-L] and the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Lung Cancer Module [EORTC QLQ LC13]), perceived life stress (quantified by the Perceived Stress Scale), and depression (quantified by the Center for Epidemiological Studies Short Depression Scale [CESD-10]), in lung cancer patients in the intervention and control conditions (control arm closed to accrual as of 3/6/2012) from baseline to 3-months following randomization.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I (closed to accrual as of 3/6/2012): Patients receive a personalized letter from their physician with advice to quit smoking and a copy of the National Cancer Institute's "Cleaning the Air" smoking cessation booklet.

ARM II: Patients receive a personalized letter and a smoking cessation booklet. Patients also receive an 8-week supply of nicotine replacement patches and undergo a counseling session over 30-45 minutes with a trained nurse or midlevel provider that focuses on the benefits of quitting smoking for cancer patients and addresses cancer-specific concerns about smoking cessation. Patients also undergo a quitline-based smoking cessation intervention comprising 5 individual 25- to 30-minute telephone counseling sessions and unlimited inbound phone-based access to Quit Coaches over 8-11 weeks, mailed written materials, and an interactive online program.

After completion of study treatment, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with American Joint Committee on Cancer (AJCC) stage I-IIIa/b non-small cell lung cancer or limited stage small cell lung cancer Smoked any cigarettes in the past seven days Willing to consider quitting smoking

Exclusion Criteria:

Patients with drug and alcohol abuse:

* All patients will be assessed for alcohol use using a validated 1-item screening question; if positive, patients will be assessed using the validated Alcohol Use Disorders Identification Test (AUDIT) screening instrument, those with scores >= 8 (the validated cutoff) will be excluded
* All patients will be assessed for drug use using a 1-item screening question: "How many times in the past month have you used an illegal drug or used a prescription medication for non-medical reasons?"; those with a response of >= 1 will be excluded Patient is unable to comprehend study documents and provide informed consent or Eastern Cooperative Oncology Group (ECOG) performance status is greater than two Patient does not read or understand English Patient refuses to participate Patient is contraindicated to receive nicotine replacement therapy: a) Patient is pregnant or breastfeeding, b) Patient has unstable cardiac disease within the past month (defined as unstable angina, myocardial infarction, serious arrhythmias, or any cardiac intervention procedure), or c) Patient is currently taking Chantix Patient does not have regular access to a phone to receive calls from the quitline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Participation of patients with lunch cancer in the outpatient oncology setting | 1 year
  Participation rate will be calculated as the proportion of the eligible patients who agree to participate.
Accrual of patients with lung cancer in the outpatient oncology setting | Over 1 year
  Estimated as the number of patients accrued divided by the number of months of accrual.
Participant retention | 3 months
  Estimated as the proportion of participating patients who complete questionnaires at the three month follow-up. Participants who discontinue the intervention but complete the outcome assessments will be counted in the numerator for calculating retention. Retention estimates will be calculated overall and by intervention arm. A Fisher exact test will be used to assess the difference in retention between the two arms. Kaplan-Meier methods will be used to estimate the time to drop-out, and a logrank test will be used to assess the difference in these distributions between treatment arms.
Participant acceptance of the enhanced quitline-based smoking cessation intervention | 3 months
  Evaluated by summarizing the intervention participants' ratings of how much they liked and found the intervention and the interventionists to be helpful and sensitive to their concerns. Exact 95% confidence intervals (CI) will be calculated for these estimates. Open-ended questions regarding these issues will be summarized using qualitative methods.
Protocol fidelity | 3 months
  Summarized by calculating the proportion of participants in both groups who report that they received advice from their physician to quit smoking, estimating the frequency with which intervention participants completed calls and calculating the mean duration of each call, and calculating the proportion of participants that utilized web-based services (including the frequency of the number of logins and sections visited and mean duration of visit).

SECONDARY OUTCOMES:
Abstinence rate in both groups | 3 months
Comparison of changes in quality of life, stress, and depressive symptoms between groups | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Weaver, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States